CLINICAL TRIAL: NCT05847985
Title: Language and Lewy Body Diseases: Sentence Comprehension Problems and Modifying Noninvasive Brain Stimulation Treatment
Acronym: LANG-LBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NU23J-04-00005
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Lewy Body Disease; Healthy Aging
MeSH Terms: conditions — Lewy Body Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Differences between LBDs patients and HC in regulation of language functions (No Intervention): In this study, 25 LBDs patients and 25 HC will undergo neuropsychological assessment, speech and writing recording, and MRI (structural T1 sequences, sentence comprehension fMRI task, neuromelanin-sensitive MRI sequence, and resting state measurement). The HC group will be matched to the LBDs patients with MCI for gender and age.
- Long-term effects of repeated sessions of home-based tDCS delivered via telepractice (Experimental): The investigators will use a parallel-group, double-blinded, randomized, sham-stimulation-controlled design. Forty LBDs patients will be randomized into two parallel groups, n = 20 subjects in each arm. For the active group, the investigators will use the stimulation protocol with the anode over the left IFG (cathode over the right supraorbital area, 2mA, 20 minutes). Participants will undergo a baseline assessment (A0, as described in arm 1); 10 stimulation sessions (in a two-week period); a follow-up assessment immediately after tDCS treatment (A1), and follow-up assessments 8 weeks (A2) after the baseline assessment. Each assessment will consist of a brief neuropsychological assessment, speech and writing recording and MRI scanning.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS using electric currents to modulate underlying neurons
  Arms: Long-term effects of repeated sessions of home-based tDCS delivered via telepractice

SUMMARY:
Lewy body diseases (LBDs) represents a group of neurodegenerative disorders characterized by the abnormal accumulation of aggregates of α-synuclein protein leading to the formation of Lewy bodies (LB) and Lewy neurites resulting in cell death. LBDs consists of two major clinical entities - Parkinson's disease (PD) and dementia with LB (DLB). Vast majority of patients with LBDs either already have mild cognitive impairment (MCI) at the time of the diagnosis or will develop it during the course of the disease. Language dysfunctions in LBDs patients with MCI are often unrecognized, which are difficult to treat, but even subtle changes might lead to impairment of social and occupational functioning with profound effect on their quality of lives. Current pharmacological or surgical strategies are effective for tackling the motor issues of LBDs with very limited effects on other symptoms such as language dysfunctions. Therefore, non-pharmacological approaches are gaining more attention. One of these non-pharmacological strategies is the use of noninvasive brain stimulation (NIBS) techniques that are able to modulate the brain functions with the effects on human nervous system plasticity. In this proposed project the investigators aim to first describe specific alterations in the language domain in LBDs patients with MCI as compared to healthy controls (HC) and identify the neural underpinnings of these changes using novel combination of advanced multimodal imaging techniques and various analytical methods. Secondly, the investigators aim to use NIBS as a supervised and individualized home-based therapeutical approach to tackle the language dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* right-handedness
* Czech as their first language
* age (60-80 years)
* presence of PD-MCI (Litvan et al. 2012) or MCI-LB (McKeith et al. 2020) for LBD subjects

Exclusion Criteria:

* cardio pacemaker
* any MRI-incompatible metal in the body
* epilepsy
* any diagnosed psychiatric disorders
* alcohol/drug abuse
* for HC group the presence of LBDs or other neurodegenerative disorder or MCI/dementia

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
sentence comprehension performance - accuracy | through study completion, an average of 1 year
  the investigators will study comprehension of syntactically complex sentences - accuracy in sentence comprehension task
sentence comprehension performance - reaction times | through study completion, an average of 1 year
  the investigators will study comprehension of syntactically complex sentences - reaction times in sentence comprehension task

SECONDARY OUTCOMES:
relation of sentence comprehension performance to cognitive performance | through study completion, an average of 1 year
  the investigators will correlate sentence comprehension with cognitive functions: z-scores in following domains - memory, attention, executive function, visuospatial function and language function of Short Neuropsychological Battery (Bolcekova et al. 2020)
The neural underpinning of sentence comprehension deficits - sentence comprehension fMRI task data | through study completion, an average of 1 year
  The investigators will identify connectivity differences between HC and LBDs patients with MCI in language-related domain-specific and domain-general networks. In the task-based fMRI study, LBDs patients with MCI will show reduced activation and altered functional connectivity within and between these large-scale cortical networks compared to HC.
The neural underpinning of sentence comprehension deficits - resting state data | through study completion, an average of 1 year
  Abnormal intra- and inter-network dynamics will be apparent in resting-state fMRI of LBDs patients with MCI as compared to HC.
The neural underpinning of sentence comprehension deficits - structural MRI data | through study completion, an average of 1 year
  LBDs patients with MCI will show structural changes in language-related domain-specific and domain-general networks with neural degeneration as assessed by NMS-MRI as compared to HC.
the long-term effects of repeated sessions of home-based tDCS on sentence comprehension - accuracy | On the beginning of the study, after completion of two-week stimulation a eight weeks after the baseline assessment
  the investigators will investigate the long-term effects of repeated sessions of home-based tDCS on sentence comprehension of syntactically complex sentences - accuracy in sentence comprehension task (as was described in outcome 1)
the long-term effects of repeated sessions of home-based tDCS on sentence comprehension - reaction times | On the beginning of the study, after completion of two-week stimulation a eight weeks after the baseline assessment
  the investigators will investigate the long-term effects of repeated sessions of home-based tDCS on sentence comprehension of syntactically complex sentences - reaction times in sentence comprehension task (as was described in outcome 2)
the long-term effects of repeated sessions of home-based tDCS on sentence comprehension - The neural underpinning of sentence comprehension deficits - resting state data | On the beginning of the study, after completion of two-week stimulation a eight weeks after the baseline assessment
  the investigators will investigate the long-term effects of repeated sessions of home-based tDCS on resting state data (as was described in outcome 5)
the long-term effects of repeated sessions of home-based tDCS on sentence comprehension - The neural underpinning of sentence comprehension deficits - sentence comprehension fMRI task data | On the beginning of the study, after completion of two-week stimulation a eight weeks after the baseline assessment
  the investigators will investigate the long-term effects of repeated sessions of home-based tDCS on sentence comprehension fMRI task data (as was described in outcome 4)
the long-term effects of repeated sessions of home-based tDCS on sentence comprehension - The neural underpinning of sentence comprehension deficits - structural MRI data | On the beginning of the study, after completion of two-week stimulation a eight weeks after the baseline assessment
  the investigators will investigate the long-term effects of repeated sessions of home-based tDCS on structural MRI data (as was described in outcome 6)

CONTACTS AND LOCATIONS:
Locations (1):
- Masaryk University CEITEC, Brno, Czechia